CLINICAL TRIAL: NCT04732364
Title: Analgesic Efficacy of Magnesium Sulphate as an Adjuvant to Levo-bupivacine in Ultrasound Guided Erector Spinae Plan Block for Modified Radical Mastectomy
Brief Title: Analgesic Efficacy of Ultrasound Guided Erector Spinae Block for Modified Radical Mastectomy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Peter Rafaat Edward Iskander, principal investigator, South Egypt Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: peter SECI
Record Dates: First submitted 2021-01-06; First posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Pain, Postoperative
Keywords: Erector Spinae Block; magnesium sulphate; dexmedetomidine
MeSH Terms: conditions — Pain, Postoperative | interventions — Mastectomy, Modified Radical; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (C) (control group): (Placebo Comparator): Patient will receive 20 ml 0.25% levobupivacaine into interfascial plane below erector spinae muscle at level of T5.
  Interventions: Procedure: ultrasound guided erector spinae plan block using bupivacaine for modified radical mastectomy
- Group (D) (Dexmetonidine group): (Active Comparator): Patient will receive 20ml 0.25% levobupivacaine + 1μ/kg dexmedetomidine into interfascial plane below erector spinae muscle at level of T5..
  Interventions: Procedure: ultrasound guided erector spinae plan block with bupivacaine and Dexmetonidine for modified radical mastectomy
- Group (M) (magnesium slphate group): (Active Comparator): Patient will receive 20ml 0.25% levobupivacaine + 0.7 mg/kg MgSo4 into interfascial plane below erector spinae muscle at level of T5..
  Interventions: Procedure: ultrasound guided erector spinae plan block with bupivacaine and magnesium slphate for modified radical mastectomy

INTERVENTIONS:
Procedure: ultrasound guided erector spinae plan block using bupivacaine for modified radical mastectomy — Ultrasound guided Erector spinae plane (ESP) block will be given with patient in sitting position depending on surgical site (left or right) ESP block will be given using high frequency linear u/s transducer, the probe is placed in longitudinal orientation lateral to thoracic fifth spinous process, then Trapezius muscle, Rhomboidus major muscle, and erector spinae muscle
  Arms: Group (C) (control group):
Procedure: ultrasound guided erector spinae plan block with bupivacaine and Dexmetonidine for modified radical mastectomy — Ultrasound guided Erector spinae plane (ESP) block will be given with patient in sitting position depending on surgical site (left or right) ESP block will be given using high frequency linear u/s transducer, the probe is placed in longitudinal orientation lateral to thoracic fifth spinous process, then Trapezius muscle, Rhomboidus major muscle, and erector spinae muscle
  Arms: Group (D) (Dexmetonidine group):
Procedure: ultrasound guided erector spinae plan block with bupivacaine and magnesium slphate for modified radical mastectomy — Ultrasound guided Erector spinae plane (ESP) block will be given with patient in sitting position depending on surgical site (left or right) ESP block will be given using high frequency linear u/s transducer, the probe is placed in longitudinal orientation lateral to thoracic fifth spinous process, then Trapezius muscle, Rhomboidus major muscle, and erector spinae muscle
  Arms: Group (M) (magnesium slphate group):

SUMMARY:
To compare the analgesic efficacy of dexmedetomidine and magnesium sulphate as adjuvants to levobupivacaine in erector spinae plane block in modified radical mastectomy surgery for acute and chronic pain management.

DETAILED DESCRIPTION:
3 groups.

Group (C) / (I):20 patient (control group) :

Patients will receive 20 ml 0.25% levobupivacaine into the interfascial plane below erector spinae muscle at level of T5.

Group (D)/ (II) :20 patient (Dexmetonidine group) :

Patient will receive 20ml 0.25% levobupivacaineas above + 1μ/kg dexmedetomidine.

Group (M) / (III) : 20 patient (magnesium slphate group) :

Patient will receive 20ml 0.25% levobupivacaineas above + 0.7 mg/kg MgSo4 . The patient, the anesthesiologist who administered the drugs, and the data collector will be blinded to the study drugs.

ELIGIBILITY:
Inclusion Criteria:

* female patient
* American society of anesthesiologists (ASA) I and II physical status
* age from 25 to 70 years old
* scheduled for either left or right modified radical mastectomy (MRM).

Exclusion Criteria:

* infection of the skin at or near site of needle puncture
* coagulopathy
* drug hypersensitivity or allergy to the studied drugs
* central or peripheral neuropathy
* significant organ dysfunction cardiac dysrrhythmias
* obesity (BMI>35kg/m2)
* recently use analgesic drugs

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-04-30 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
analgesia requirement | 24 hours
  first request for analgesia and total analgesia requirements

SECONDARY OUTCOMES:
chronic pain assessment | 6 months
  Assessment of chronic pain at 1-3 and 6 month post-operatively using LANSS pain score. a score of 12 or more is suggestive of neuropathic pain.

CONTACTS AND LOCATIONS:
Overall Officials: peter R Edward, MSc, Principal Investigator — specialist
Locations (1):
- South Egypt Cancer Institute, Asyut, Egypt